CLINICAL TRIAL: NCT02571764
Title: The Effect of Supplementary Food on Recovery From Moderate Acute Malnutrition in Pre-school Children in Rural Mexico
Brief Title: Supplementary Food for Moderate Acute Malnutrition in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-1409
Record Dates: First submitted 2015-09-29; First posted 2015-10-08 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Moderate Acute Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutritional Oats Cookie (Experimental)
  Interventions: Other: Nutritional Oats Cookie

INTERVENTIONS:
Other: Nutritional Oats Cookie

SUMMARY:
Children with moderate acute malnutrition will be recruited in order to receive an intervention which consists in the consumption of a single serving of SF-cookies daily, 7-days a week for 12 months and 12 educational sessions on health and nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Children (2-5 years old), who are from low socioeconomic classes (E and D classes),
* reside in rural areas, and with WHZ- between > -3 and ≤ -2, and
* informed consent given by the subject's mother or caregiver

Exclusion Criteria:

* Severe acute malnutrition (HAZ, WAZ and WHZ-scores ≤-3) based on the 2006 World Health Organization (WHO) reference values (24)
* Vitamin A deficiency (softening, ulceration, cloudiness of the cornea, and dryness of the conjunctivitis), and iodine deficiency (visible goiter)
* (3 or more episodes of loose/liquid stools/per day and lasted more than 24-hours), fever (high temperature that lasted more than 24 hours as reported by the mother/caregiver), and respiratory infections (coughing and/or runny nose that last more than 24 hours).
* Current consumption of other supplementary foods.
* Peanut or other ingredient allergy based on prior report. If some direct family member is allergic to peanuts, child would not be enrolled.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 248 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Weight (kg) for height (cm) Z-score | 12 months

SECONDARY OUTCOMES:
Weight (kg) gains | 12 months
height (cm) for age (months) Z-score | 12 months
weight (kg) for age (months) Z-score | 12 months
Mid-upper arm circumference (cm) (MUAC) | 12 hours
height (cm) gain | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Juan Osvaldo Talavera Piña, PhD, Principal Investigator — Universidad Autónoma del Estado de México
Locations (1):
- Un Kilo de Ayuda, Colonia Lomas de Chapultepec, Mexico City, Mexico